CLINICAL TRIAL: NCT01630174
Title: Phase I Study of Concurrent Selective Lymph Node Late Course Accelerated Hyper-fractionated Radiotherapy and Pemetrexed, Cisplatin for Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: IMRT/Pemetrexed/Cisplatin in Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Baosheng Li, Ph.D., Shandong Cancer Hospital and Institute
Other Study IDs: phase 1 pem IMRT
Record Dates: First submitted 2012-06-27; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Esophageal Cancer
Keywords: IMRT,Pemetrexed,Cisplatin , Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate the effect of concomitant late course accelerated hyperfractionation radiochemotherapy with pemetrexed and cisplatin in patients with esophagus cancer

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent; 2.Acquired pathological diagnosis; 3.Life expectancy≥6 months; 4.Age:18-75 years, male or female; 5.General state of health: ECOG 0-1 grade; 6.Without any chemotherapy or radiotherapy; 7.Subjects meet the following criteria for the clinical laboratory:HG≥100g/L, WBC≥3.5X109 /L, neutrophilic leukocyte≥1.5X109,PLT100X109 /L。CR≤1.5 x N，TB≤2.5XN，AST and ALT≤2.5xN，AKP≤2.5XN.

Exclusion Criteria:

* 1.Serious infection; 2.Uncontrollable diabetes; 3.Other serious diseases, such as myocardial infarction in 6 months; 4. Participated other clinical trials in 4 weeks or at present

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: esophagus cancer patients
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-10

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer hospital and institute, Jinan, Shandong, China